CLINICAL TRIAL: NCT04108715
Title: Erector Spina Plane Block Versus Deep Serratus Anterior Plane Block for Post Mastectomy Analgesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Saud University (Other)
Responsible Party: Principal Investigator, Ahmed Khaled Thallaj, Associate professor, King Saud University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: E-19-3943
Record Dates: First submitted 2019-07-07; First posted 2019-09-30 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: MASTECTOMY

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor is not aware of the study type
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ESPB GROUP (Active Comparator): Erector spina plane block group
  Interventions: Procedure: Erector spina plain block for mastectomy analgesia
- SAPB group (Active Comparator): Deep Serratus anterior plane block group
  Interventions: Procedure: Deep serratus anterior plane block

INTERVENTIONS:
Procedure: Erector spina plain block for mastectomy analgesia — After giving general anesthesia, patient is positioned in lateral decubitus with the surgical side up, An erector Spina plain block is performed with inserting block needle (Pajunk, Geisingen, Germany) in-plane under ultrasound control until needle tip hits the transverse process, a volume of 0.3 ml/kg of bupivacaine 0.25% (Marcaine, Astra Zeneca Pharmaceuticals) is injected. Pain management assessment and analgesic consumption will be provided through patient-controlled analgesia (PCA) for 24 hours. The PCA pump is programmed to deliver 1 mg morphine bolus per press with a lockout interval of 10 min. Pain scores will be measured using eleven points numerical rating scale NRS (0 to 10) and opioids consumption will be documented at 0, 1, 4, 8 and 24 hours. Time of admission to post-anesthesia care unit PACU is considered 0 hours. Any opioid equivalents given during the first 24 hours to manage breakthrough pain will be documented
  Arms: ESPB GROUP
Procedure: Deep serratus anterior plane block — After giving general anesthesia, the patient is positioned in lateral decubitus, with the surgical side up. The upper arm is abducted and elevated above the head level. A block needle is introduced in-plane, targeting the plane deep to the serratus anterior muscle, and a bolus of 0.3 ml/kg bupivacaine 0.25% is injected through ultrasound guidance. Pain management assessment and analgesic consumption will be provided through patient-controlled analgesia PCA for 24 hours. The PCA pump is programmed to deliver 1 mg morphine bolus per press with a lockout interval of 10 min. Pain scores will be measured using eleven points numerical rating scale NRS (0 to 10), and opioids consumption will be documented at 0, 1, 4, 8 and 24 hours. Time of admission to PACU is considered 0 hours. Any opioid equivalents given during the first 24 hours to manage breakthrough pain will be documented
  Arms: SAPB group

SUMMARY:
Breast cancer surgery like Mastectomy and modified radical mastectomy are associated with significant postoperative pain, and management depends largely on patient controlled analgesia with intravenous Morphine or other opioids equivalents. Respiratory depression, Ileus, sedation, nausea and vomiting are some of the potential side effect of opioid treatment which prolonged hospital length of stay and increase the coast. Recent advance in ultrasound guided regional anesthesia has led to the development of two novel regional anesthesia techniques specific to chest wall analgesia; Erector spina plain block and Serratus anterior plain block, with its potential to reduce or eliminate the need for opioids to manage post-operative pain.

DETAILED DESCRIPTION:
Experimental: erector spinae plain block After giving general anesthesia, patient is positioned in lateral decubitus with the surgical side up, and prepping para-spinous area with antiseptic solution. Ultrasound high frequency linear transducer is positioned in a para-sagittal plane at the level of fifth thoracic vertebra. Scanning of interested structures from superficial to deep planes, Trapezius muscle, Rhomboid major muscle, Erector spina muscle and transverse process of fifth thoracic vertebra.

Comparator: serratus anterior plane block After giving general anesthesia, patient is positioned in lateral decubitus, with the surgical side up. The upper arm is abducted and elevated above the head level. Under sterile aseptic technique, a linear ultrasound transducer (6-15 MHz) is placed in a sagittal oblique plane over the fourth and fifth ribs at the mid-axillary line. The following muscles are identified overlying the fourth/ fifth rib: the latissimus dorsi (superficial) and serratus anterior muscle (deep) overlying the ribs.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III patients age 18 to 75 years undergoing unilateral breast surgery

Exclusion Criteria:

* Patients refusal
* History of amide local anesthetics allergy
* Alcohol or drug abuse
* Chronic opioid intake
* Language barriers
* Patient with psychiatric disorders
* Contraindications for regional anesthesia
* BMI > 40 Kg/m2
* Obstructive sleep apnea that preclude PCA opioids

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2019-07-07 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-26 (Actual)

PRIMARY OUTCOMES:
Cumulative Opioid consumption in the first 24 hours. | 0 hours post- operative( 0 time is considered time to admission to post anesthesia care unit)
  Post- operative morphine consumption measured from patient controlled analgesia pump (PCA machine)
Cumulative Opioid consumption in the first 24 hours. | 1 hour post-operative
  Post- operative morphine consumption measured from patient controlled analgesia pump (PCA machine)
Cumulative Opioid consumption in the first 24 hours. | 4 hours post-operative
  Post- operative morphine consumption measured from patient controlled analgesia pump (PCA machine)
Cumulative Opioid consumption in the first 24 hours. | 8 hours post-operative
  Post- operative morphine consumption measured from patient controlled analgesia pump (PCA machine)
Cumulative Opioid consumption in the first 24 hours. | 24 hours post-operative
  Post- operative morphine consumption measured from patient controlled analgesia pump (PCA machine)
Post-operative pain intensity | pain at 0 hour, 0 time is considered time to admission to post anesthesia care unit
  pain intensity is measured by ( 11 point numerical scale from 0 to 10), where 0 is considered no pain, 10 is the worst pain
Post-operative pain intensity | pain at 1 hour post operative
  pain intensity is measured by ( 11 point numerical scale from 0 to 10), where 0 is considered no pain, 10 is the worst pain
Post-operative pain intensity | pain at 4 hours post operative
  pain intensity is measured by ( 11 point numerical scale from 0 to 10), where 0 is considered no pain, 10 is the worst pain
Post-operative pain intensity | pain at 8 hours post operative
  pain intensity is measured by ( 11 point numerical scale from 0 to 10), where 0 is considered no pain, 10 is the worst pain
Post-operative pain intensity | pain at 24 hours post operative
  pain intensity is measured by ( 11 point numerical scale from 0 to 10), where 0 is considered no pain, 10 is the worst pain

SECONDARY OUTCOMES:
Time to patient mobilization | First 24 hours post operative( 0 time is considered time to admission to post anesthesia care unit)
  Recording first time patient is able to mobilize without assistance

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Thallaj, Principal Investigator — King Saud University
Locations (1):
- King Saud University, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No